CLINICAL TRIAL: NCT04981899
Title: Multicenter Study of Safety and Efficacy of PET-adapted Treatment With Nivolumab at the Fixed Dose 40 mg, Ifosfamide, Carboplatin, Etoposide (NICE-40) in Patients With Relapsed/Refractory Hodgkin Lymphoma
Brief Title: A Study of Safety and Efficacy of PET-adapted Treatment With Nivolumab at the Fixed Dose 40 mg, Ifosfamide, Carboplatin, Etoposide (NICE-40) in Patients With Relapsed/Refractory Hodgkin Lymphoma
Acronym: NICE-40
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: r/r cHL NICE-40
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Nivolumab; Ifosfamide; Carboplatin; Etoposide
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main arm (Experimental): Patients will receive 6 cycles of nivolumab at the fixed dose of 40 mg, with subsequent assessment of response by PET-CT. Patients with CR will proceed to ASCT.
  Patients with <CR after nivolumab monotherapy will be treated with 2 cycles of a combination of nivolumab at the fixed dose 40 mg, ifosfamide, carboplatin and etoposide (NICE-40), with subsequent PET-CT assessment.
  Interventions: Drug: Nivolumab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Nivolumab — 6 infusions of nivolumab at a fixed dose of 40 mg, 14 days apart, and infusion of nivolumab on day 0 of the NICE-40.
Drug: Ifosfamide — 5000 mg / m2, 24-hour infusion on day 2 of the NICE-40.
Drug: Carboplatin — Optimized to get AUC = 5 (max. 800 mg) on day 2 of the NICE-40.
Drug: Etoposide — 100 mg / m2 intravenously on 1-3 days of the NICE-40.

SUMMARY:
Nivolumab is an anti-PD-1 antibody highly effective in patients with relapsed/refractory classical Hodgkin lymphoma. A PET-adapted regimen of Nivo combined with ICE as first salvage therapy was shown to induce high response rates and favorable progression-free survival as a bridge to autologous stem cell transplantation, allowing to omit salvage chemotherapy in a substantial proportion of r\r cHL patients. This study evaluates the safety and efficacy of PET-adapted treatment of nivolumab at the fixed dose of 40 mg in combination with ifosfamide, carboplatin, and etoposide (NICE-40) in patients with relapsed/refractory Hodgkin Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed Hodgkins lymphoma
* Relapsed or refractory disease after the first line of treatment
* Age 18-70 years old
* Ejection fraction greater than 50%
* ECOG 0-2 status
* Signed informed consent
* No severe concurrent illness

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Severe organ failure: creatinine more than 2 norms; ALT, AST more than 5 norms; bilirubin more than 1.5 norms
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign an informed consent
* Active or prior documented autoimmune disease requiring systemic treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | 12 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).
Overall Response Rate (ORR) | 12 months
  Overall response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by LYRIC and Lugano 2014 criteria

SECONDARY OUTCOMES:
Duration of Response (DOR) | 24 months
Overall Survival (OS) | 24 months
Progression-Free Survival (PFS) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kulagin, MD,PhD, Study Director — RM Gorbacheva Research Institute of Pediatric Oncology, Hematology and Transplantation, Pavlov University
Locations (3):
- Russia (3):
  - National Medicine Research Center of oncology named after N.N. Petrov, Saint Petersburg, Pesochny
  - Irkutsk Regional Cancer Center, Irkutsk
  - St. Petersburg State Pavlov Medical University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided